CLINICAL TRIAL: NCT06762730
Title: A Single Dose Intravenous Administration of Zoledronic Acid for the Prevention of TDF-sparing ART-induced Bone Mass Density Loss in Treatment-naive HIV Positive Individuals - a Prospective, Multicenter, Open-label, Randomized Control Trial
Brief Title: Zoledronic Acid for the Prevention of TDF-sparing ART-induced Bone Mass Density Loss in Treatment-naive HIV Positive Individuals
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Sheba Medical Center (Other Government); Rambam Hospital, Haifa, Israel (Unknown)
Responsible Party: Principal Investigator, Hila Elinav, Professor, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012724-HMO-CTIL
Record Dates: First submitted 2024-12-31; First posted 2025-01-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2024-12

CONDITIONS: HIV Infected Individuals; Osteopenia
Keywords: Osteopenia; zoledronic acid; HIV naïve
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Zoledronic acid (Experimental): Patients with T score from -1 to -2.4 will be treated with 1 dose of 5 mg of Zoledronic acid within a month of ART intiation.
  Interventions: Drug: Zoledronic Acid 5 mg/Bag 100 ml Inj
- Follow up-comparator (No Intervention): Patients with T score from -1 to -2.4 that will be followed without intervention
- mildly osteopenic patients (No Intervention): patients with T score more than -1 will be followed only after antiviral treatment initiation- P1NP and CTX levels and DXA up to 4 years
- Osteoporotic patients (No Intervention): patients with T score less than -2.5 will be treated according to standard of care with oral biphosphonates, and will be followed after antiviral treatment intiation- P1NP + CTX and DXA up to 4 years

INTERVENTIONS:
Drug: Zoledronic Acid 5 mg/Bag 100 ml Inj — Zolendric acid will be provided to HIV naïve patients with documented osteopnia
  Arms: Zoledronic acid

SUMMARY:
The goal of this clinical trial is to learn if zolendric acid can prevent the anticipated deterioration of bone mass after antiviral treatment initiation for people that were recently diagnosed with HIV.

The main questions it aims to answer are:

1. Is bone mass deterioration is significant even with the new medication currently used to treat HIV?
2. Can one dose of Zolendric acid protect from deterioration of bone mass.

Researchers will compare one dose of zolendric acid to follow-up only

Participant will:

1. Provide blood samples for bone markers before antiviral treatment initiation and at 6M,12M,24M and 48M after treatment initiation
2. Perform DXA scan soon after antiviral treatment initiation and after 12M ,24 M and 48 months
3. Half of the patients with moderate reduction in bone mass will be treated with one dose of zolendric acid in the clinical trial, the other participants will be followed without intervention.
4. Patients with substantial osteoporosis will be treated according to standard of care by their HMO, but will continue followup in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age of 18 years old of any gender, social, religious or racial background.
* Confirmed positive result for HIV infection.

Exclusion Criteria:

Patients who received previous pharmacological agents for the prevention of HIV infection.

* Women who are pregnant, lactating or those who plan to become pregnant within the trial timeframe.
* Past history of severe drug-induced reaction (including atypical femur fractures or osteonecrosis of the jaw) or documented hypersensitivity to a bisphosphanate agent.
* Patients with untreated hypocalcemia at screening.
* Severe dental status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone density at 12 months. | 12 months of initiation of ART
  Average change (in %) from baseline in spine T score and hip T-score values among participants in the intervention group versus participants in the control group at 12 months after ART initiation

SECONDARY OUTCOMES:
Bone density at 24 months. | 24 months
  Average change (in %) from baseline in spine T score and hip T-score values among participants in the intervention group versus participants in the control group at 24. ART.
Bone density at 48 months. | 48 months of initiation of ART
  Average change (in %) from baseline in spine- and hip T-score values among participants in the intervention group versus participants in the control group at 48 months of initiation of ART.
Bone fractures at 48 months | 48 months of initiation of ART
  To estimate the rates of clinical fractures among all participants over a minimum of 48 months and the difference, if any, between treatment arms.
Bone markers differences during folloe up | 6,12,24,48 months after treatment intiation
  Identify difference in average blood levels of bone turnover markers between treatment arm and the non intervention arm during the follow-up period.
BMD decline in TDF sparing ART | 48 months of initiation of ART
  Rates of BMD decline (by means of rate of naïve PLHIV with baseline T score > -1.0 who will turn to T score <-1.0) in PLHIV treated with TDF-sparing ART over a period of 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hila Elinav, Doctor, Principal Investigator — Hadassah University Medical center; Eynat Kedem, Doctor, Principal Investigator — Rambam Health Care Campus; Itzchak Levy, Proffesor, Principal Investigator — Sheba Medical Center
Locations (3):
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: Undecided